CLINICAL TRIAL: NCT07317583
Title: Improving 5-Fluorouracil (5-FU) Continuous Infusion Comfort With a New Corset Design in People Affected by Cancer: A Feasibility Study
Brief Title: Improving 5-Fluorouracil (5-FU) Continuous Infusion Comfort With a New Corset Design in People Affected by Cancer
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, EZGI BILMIC, Nurse Specialist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-19-09
Record Dates: First submitted 2025-11-30; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; 5-Fluorouracil (5-FU)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group, randomized controlled feasibility trial designed to evaluate the effectiveness and usability of a newly developed supportive corset for patients receiving continuous 5-Fluorouracil (5-FU) infusion therapy. Forty colorectal cancer patients were randomly assigned to two groups: an intervention group using the corset in addition to standard care and a control group receiving standard care only. The intervention lasted four weeks, and outcomes were assessed at baseline and post-intervention using the Visual Analog Scale (VAS) for infusion-related experiences and the EORTC QLQ-C30 for quality of life.
Masking Description: This study is open-label; no masking was applied. Both participants and researchers were aware of group assignments because the intervention involved the use of a visible supportive corset during continuous 5-FU infusion therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Supportive Corset (Experimental): Participants receive standard care plus a specially designed supportive corset during continuous 5-FU infusion.
  Interventions: Device: Supportive Corset
- Standard of Care (Other): Participants receive routine care without any additional intervention.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Supportive Corset — A specially designed supportive corset developed to stabilize the 5-FU infusion pump and serum set during continuous infusion therapy. It includes a body-wrapping belt, adjustable shoulder strap aligned with the port catheter, and a fluid-proof pouch for carrying the infusion pump. The corset aims to enhance comfort, reduce physical and psychological distress, and improve overall treatment experience.
  Arms: Standard of Care + Supportive Corset
Other: Standard care — Routine care provided during continuous 5-FU infusion without any additional supportive device.
  Arms: Standard of Care

SUMMARY:
This feasibility randomized controlled trial aims to evaluate the effectiveness and usability of a newly designed supportive corset for patients receiving continuous 5-Fluorouracil (5-FU) infusion therapy. The corset is intended to stabilize the infusion pump and serum set, reduce physical and psychological discomfort, and improve overall quality of life. Forty colorectal cancer patients were randomized into two groups: an intervention group using the corset and a control group receiving standard care. Outcomes include infusion-related experiences (measured by Visual Analog Scale) and quality of life (assessed by EORTC QLQ-C30).

DETAILED DESCRIPTION:
Continuous infusion of 5-Fluorouracil (5-FU) via portable pumps is a common treatment modality for colorectal cancer, offering clinical benefits such as stable plasma drug levels and improved tolerability. However, patients often experience physical discomfort, restricted mobility, sleep disturbances, anxiety, and aesthetic concerns related to the infusion pump. Technical issues such as unstable connections and medication flow interruptions may further compromise treatment safety.

To address these challenges, this study introduces a newly designed supportive corset aimed at stabilizing the infusion pump and serum set during continuous 5-FU therapy. The corset is designed to enhance comfort, reduce movement-related anxiety, and improve sleep quality and overall treatment experience. This feasibility trial enrolled 40 patients diagnosed with colorectal cancer from an outpatient chemotherapy unit in Türkiye. Participants were randomized into two groups: the intervention group received the corset in addition to standard care, while the control group received standard care only.

Data were collected at baseline and after four weeks using the Visual Analog Scale (VAS) for infusion-related experiences and the EORTC QLQ-C30 for quality of life. The primary outcomes include changes in physical restrictions, insomnia, anxiety during movement, aesthetic concerns, and overall quality of life. Secondary outcomes include patient satisfaction with the corset. The study was approved by the Clinical Research Ethics Committee (Approval No: 2023-19-09) and conducted in accordance with ethical standards. Findings will inform the feasibility and potential integration of supportive physical devices into cancer care protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer
* Currently receiving chemotherapy
* Having received at least one cycle of 5-FU therapy via continuous infusion
* Volunteering to participate in the study
* Aged 18 years or older

Exclusion Criteria:

* Diagnosis of brain cancer (excluded due to potential impact on cognitive function and reliability of self-reported data)
* Presence of bone metastases
* Pregnancy and/or lactation
* Communication barriers
* Physician-diagnosed mental illness
* Inability to speak or understand Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Physical Restrictions Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.
Insomnia Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.
Anxiety During Movement Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.
Skin Contact Discomfort Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.
Medication Flow Issues Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.
Aesthetic Concerns Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.
Nausea Score (Visual Analog Scale) | 4 weeks
  Assessed using Visual Analog Scale (0 = never experienced, 10 = experienced very frequently). Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Quality of Life Score (EORTC QLQ-C30) | 4 weeks
  Assessed using EORTC QLQ-C30 questionnaire (30 items). Functional scales: higher scores = better functioning; symptom scales: higher scores = worse symptoms. Range: 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan Bağçivan, PHD, Study Director — University of Massachusetts Dartmouth, North Dartmouth, United States, Department of Adult Nursing, College of Nursing and Health Sciences
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Bakirköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No